CLINICAL TRIAL: NCT03310346
Title: Prospective Multicenter Registry for Preterm Newborns With Severe Pulmonary Hypertension
Brief Title: Registry of Preterm Newborns With Severe Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-2491
Record Dates: First submitted 2017-09-15; First posted 2017-10-16 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Pulmonary Hypertension; Preterm Infant
MeSH Terms: conditions — Hypertension, Pulmonary; Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this prospective research registry is to collect data on treatment strategies and outcomes for premature newborns with severe pulmonary hypertension (PH).

DETAILED DESCRIPTION:
There is a lack of consensus on the role of inhaled nitric oxide (iNO) therapy and other pulmonary vasodilators for the treatment of severe pulmonary hypertension (PH) in premature newborns (<34 weeks gestation). However, a proper randomized, controlled trial of iNO in premature newborns with severe PH has not been completed. Some practices embrace the American Academy of Pediatrics (AAP) statement that there is no condition for which iNO should be used in the premature newborn, and others selectively treat premature infants with inhaled nitric oxide (iNO) who suffer life threatening hypoxemia due to suprasystemic PH and right-to-left veno-arterial admixture across the arterial duct and/or oval foramen. The number of neonatal intensive care units (NICUs) adopting each of these approaches is currently unknown, but it is possible that the former group is increasing due to administrative pressure to reduce uncompensated off-label iNO use. A prospective registry collection of treatment strategies and outcomes for this subset of premature newborns will help define current treatment strategies and yield important information about safety and efficacy of the different approaches to management, and would inform the debate more effectively than a series of iNO treated infants alone. Data collected includes maternal age, race/ethnicity, pregnancy and delivery complications, prenatal medications, infant characteristics such as Apgar scores, birthweight, congenital anomalies, respiratory status, pharmacologic therapy used for PH and its side effects, and blood gas data. Up to 100 sites in North America will be invited to monitor for appropriate cases.

ELIGIBILITY:
Inclusion Criteria:

* Premature newborns 23-34 weeks gestation
* Echocardiographic evidence showing systemic or suprasystemic levels of PH, or > 5% difference in pre-post ductal saturation if echo is not available.
* Fraction of inspired oxygen (FiO2) >0.60 in the first 72 hours after birth

Exclusion Criteria:

* None

Ages: 0 Minutes to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Premature newborns and their mothers recruited from up to 100 neonatal intensive care units
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-07-02 (Actual); Study Completion 2022-07-02 (Actual)

PRIMARY OUTCOMES:
Mortality | From birth through hospital discharge or death, whichever occurs first, assessed up to one year
  Occurrence of death
Cause of death | From birth through hospital discharge or death, whichever occurs first, assessed up to one year
  The cause, if death occurred

SECONDARY OUTCOMES:
Number of Days Hospitalized | From birth through hospital discharge or death, whichever occurs first, assessed up to one year
  Total number of days in hospital
Number of Days on Ventilation | From birth through hospital discharge or death, whichever occurs first, assessed up to one year
  Total number of days on mechanical ventilation
Classification of Bronchopulmonary Dysplasia (BPD) | At 36 weeks after birth
  BPD classification
Development of Necrotizing Enterocolitis (NEC) | From birth through surgical repair of NEC, assessed up to one year
  Occurrence of surgical repair of NEC
Development of Early Bacterial Sepsis | From Birth through 3 days of life
  Early Occurrence of Bacterial sepsis, e.g. 3 days or less
Development of Late Bacterial Sepsis | From Day 4 of life through hospital discharge or death, whichever occurs first, assessed up to one year
  Late Occurrence of Bacterial sepsis, e.g. >3 days
Intracranial hemorrhage | From birth through hospital discharge or death, whichever occurs first, assessed up to one year
  Occurrence and severity of intracranial hemorrhage
Cystic Periventricular Leukomalacia (PVL) | From birth through hospital discharge or death, whichever occurs first, assessed up to one year
  Occurrence of PVL
Surgery for Retinopathy of Prematurity (ROP) | From birth through hospital discharge or death, whichever occurs first, assessed up to one year
  Occurrence of surgical repair of ROP
Patent Ductus Arteriosus (PDA) Ligation | From birth through hospital discharge or death, whichever occurs first, assessed up to one year
  Occurrence of surgical repair of PDA
Pneumothorax | From birth through hospital discharge or death, whichever occurs first, assessed up to one year
  Occurrence of pneumothorax
Neurological Exam | The most recent exam immediately prior to discharge or death, whichever occurs first, assessed up to one year
  Results of neurological exam: Normal, Abnormal, Suspect

CONTACTS AND LOCATIONS:
Overall Officials: John P Kinsella, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No